CLINICAL TRIAL: NCT00211978
Title: EPIC (Effect of PhosLo on Phosphorus Levels in Chronic Kidney Disease): A Prospective, Multicenter, Randomized, Double-Blinded, Placebo-Controlled, Parallel Arm, Study of PhosLo on Phosphorus Levels in Subjects With Chronic Kidney Disease
Brief Title: EPIC(Effect of PhosLo on Phosphorus Levels in Chronic Kidney Disease)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Responsible Party: Paul Kessler, MD, Sr. VP, Clinical, Medical, & Regulatory Affairs, Nabi Biopharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nabi 6402; EUDRACT# 2005-002565-36
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-12

CONDITIONS: Hyperphosphatemia; Kidney Failure
Keywords: PhosLo (Calcium acetate)
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency | interventions — calcium acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PhosLo (Experimental)
  Interventions: Drug: calcium acetate
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: calcium acetate — 667 mg gelcaps, 1-3 t.i.d. (titrated to serum phosphorus level)
  Other Names: PhosLo
  Arms: PhosLo
Drug: placebo — gelcap, 1-3 t.i.d. (titrated to serum phosphorus level)
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if calcium acetate (PhosLo) can control serum phosphorus in pre-dialysis patients with moderate to severe impairment of kidney function.

DETAILED DESCRIPTION:
In patients with impaired kidney function, dietary phosphorus can not be completely excreted, which leads to elevated levels of serum phosphorus. Elevated serum phosphorus leads to increased levels of parathyroid hormone (PTH), and is associated with bone disease and other adverse consequences such as soft-tissue and vascular calcification, and increased morbidity and mortality. It is therefore important to prevent hyperphosphatemia and maintain serum phosphorus levels within the range recommended by K/DOQI. In patients on dialysis, phosphate binders are routinely used to control serum phosphorus by absorbing dietary phosphate during the transit through the intestine. However, the use of phosphate binders for non-dialyzed patients with chronic kidney disease (CKD) is not an FDA approved indication, although some physicians treat patients prior to dialysis based on clinical judgment. The goal of this study is to demonstrate the efficacy of calcium acetate (PhosLo) in controlling serum phosphorus in patients with moderate to severe decrease in kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Non-dialyzed male or female patients with CKD, with a GFR of less than 30mL/min/1.73m² who have elevated serum phosphorus or who develop elevated serum phosphorus following washout from phosphorus-binding therapy.
* Patients must have written informed consent
* Negative serum pregnancy test if appropriate
* Expected to be able to comply with protocol procedures and schedule

Exclusion Criteria:

* Unstable angina pectoris
* Severe congestive heart failure
* Severe liver dysfunction
* Severe malnutrition
* Severe hyperparathyroidism
* AIDS (HIV positive subjects without AIDS are not excluded)
* Active malignancy for which the subject is receiving chemotherapy or radiation
* Subject unlikely to complete the study
* History of obstructed bowels or hypersensitivity to any of the study medications or their components
* History of swallowing disorders such as dysphagia (that would prevent the subject from taking the study drug) severe gastrointestinal motility disorders, or major GI tract surgery
* Participation in an investigational drug or device trial within 30 days of randomization
* Subjects on Vitamin D therapy
* Subjects with acute symptoms, in the last month, or current radiographic evidence of kidney stones
* Subjects who have undergone renal transplant or receiving dialysis
* Or any condition with makes patient participation not in the patients best interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-05; Primary Completion 2006-06 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
serum phosphorus | weeks 5-24

SECONDARY OUTCOMES:
calcium x phosphorus product | weeks 5-24
intact parathyroid hormone | weeks 5-24

CONTACTS AND LOCATIONS:
Overall Officials: Wajeh Y Qunibi, M.D., Study Chair — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Sciences Center, San Antonio, Texas, United States

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Qunibi W, Winkelmayer WC, Solomon R, Moustafa M, Kessler P, Ho CH, Greenberg J, Diaz-Buxo JA. A randomized, double-blind, placebo-controlled trial of calcium acetate on serum phosphorus concentrations in patients with advanced non-dialysis-dependent chronic kidney disease. BMC Nephrol. 2011 Feb 16;12:9. doi: 10.1186/1471-2369-12-9. PMID 21324193